CLINICAL TRIAL: NCT05344586
Title: The Effects of Neural Load on Hamstring Stretching Upon Range of Motion, Maximum Isometric Strength and Tibial Nerve Pressure Pain Threshold in Asymptomatic Patients
Brief Title: The Effects of Hamstring Stretching With and Without Neural Load on Flexibility, Maximum Isometric Strength and Tibial Nerve Pressure Pain Threshold
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Alexander Achalandabaso, Principal Investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEIM/HU/2019/36
Record Dates: First submitted 2022-04-15; First posted 2022-04-25 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Hamstring stretching program with neural load
  Interventions: Other: Hamstring stretching program with neural load
- Control group (Experimental): Hamstring stretching program without neural load
  Interventions: Other: Hamstring stretching program without neural load

INTERVENTIONS:
Other: Hamstring stretching program with neural load — Participants will perform a hamstring stretch with neural load on their dominant leg. They will stretch five days a week, carrying out two repetitions of one minute each, taking a thirty second break in between. The stretch will be performed in a standing position with their dominant leg on a surface at a mid-thigh height approximately, where their knee is not fully stretched and remains unlocked and their back is in a neutral position. Participants will be encouraged to keep a maximum stretching sensation without feeling any pain. To perform the stretch, different tension parameters will be added in the following order (the next parameter shall not be introduced until the previous one has been exhausted): ankle dorsiflexion, cervical and craniocervical flexion, and hip flexion.
  Arms: Intervention group
Other: Hamstring stretching program without neural load — Participants will perform a hamstring stretch without neural load on their dominant leg. They will stretch five days a week, carrying out two repetitions of one minute each, taking a thirty second break in between. The stretch will be performed in a standing position with their dominant leg on a surface at a mid-thigh height approximately, where their knee is not fully stretched and remains unlocked and their back is in a neutral position. Participants will be encouraged to keep a maximum stretching sensation without feeling any pain. To perform the stretch, tension will be added by flexing their hip, keeping their ankle relaxed and their spine neutral.
  Arms: Control group

SUMMARY:
The study will be carried out at the Faculty of Nursing and Physiotherapy of the University of Alcala. The study has been approved by the Animal Research and Experimentation Ethics Committee of the University of Alcalá. Healthy subjects will be recruited and divided into two groups randomly to perform a hamstring stretching program for two months.

One group will perform a stretch with neural load and the other without neural load, although both groups will stretch for the same amount of time, repetitions and subjective sensation.

Participants will be measured before and after performing their assigned stretch. Then, a new post-stretch measurement will be taken after two months, period during which the subjects will perform the stretching program on their own. Finally, subjects will be asked to quit the stretching program to take a final evaluation measurement after one month of follow-up.

The objective will be to evaluate the effects of stretching with and without neural load on hamstring flexibility (main variable), maximum isometric strength and tibial nerve pressure pain threshold.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects who do not perform hamstring stretches with neural load in their daily training routine

Exclusion Criteria:

* Elite athletes competing or preparing for competition
* Lower limb surgery
* Hamstring injury in the last year
* Neurological, rheumatologic and/or orthopedic pathological history of lower limbs.
* Other comorbidities

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
Changes in hamstring flexibility | Baseline, 2 months and 3 months after intervention commencement
  measured with a goniometer. The subject remains in a supine position with both lower limbs extended. One examiner maintains a 90° hip flexion of the lower limb chosen for measurement, while the other examiner passively brings the knee to extension until a greater tissue resistance is noted or a feeling of discomfort is indicated by the subject. The knee extension is measured taking as reference the articular interline, the peroneal malleolus and the greater trochanter. The ankle remains in a relaxed position and the first examiner checks that no pelvic tilts occur while measuring.
  It is determined whether the subject has hamstring retraction if he scores less than 160º.

SECONDARY OUTCOMES:
Changes in maximum isometric hamstring strength | Baseline, 2 months and 3 months after intervention commencement
  measured using a digital dynamometer. Participants are placed in a prone position on the stretcher with the lower limb chosen for measurement in a 90º knee flexion (position determined visually). The dynamometer is placed on the subject´s heel. Then, an increasing force towards the knee extension is applied for 3-5 seconds. Subjects must try to maintain this position without allowing the knee to extend. The measurement is taken when the subject begins to extend his knee. Three measurements are taken in the same position leaving 30 seconds of rest in between. Finally, the average of the three measurements is taken.

OTHER OUTCOMES:
Changes on tibial nerve pressure pain threshold | Baseline, 2 months and 3 months after intervention commencement
  measured with a pressure algometer. Participants are placed in a prone position on the stretcher with both lower limbs extended. Measurements are taken in the popliteal fossa at the midpoint of the knee flexor line. The subject is instructed to report when pain and/or discomfort begins to be noticeable. Three different measurements are taken on the dominant leg leaving a 10 second rest in between. The pressure pain threshold value is the mean of the three measurements obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Mínguez, Principal Investigator — University of Alcalá, Madrid, Spain
Locations (1):
- Juan, Alcalá de Henares, Madrid, Spain